CLINICAL TRIAL: NCT06668857
Title: Oculomotor Profile in Acute Vestibular Syndrome - Value of Saccades, Pursuit Eye Movements and Pupillary Reflexes in Differentiating Central and Peripheral Causes
Brief Title: Quantitative Eye Movement Measurements in Patients with Acute Vestibular Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexander Tarnutzer (Other)
Responsible Party: Sponsor-Investigator, Alexander Tarnutzer, Senior leading physician, Kantonsspital Baden
Organization: Kantonsspital Baden (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Okulomotorikstudie_KSB_2024
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Acute Vestibular Syndrome; Vertigo; Stroke Acute; Acute Unilateral Vestibulopathy (AUV)
Keywords: vertigo; dizziness; acute vestibular syndrome; stroke; vestibular neuritis; diagnostic accuracy
MeSH Terms: conditions — Vertigo; Stroke; Dizziness; Vestibular Neuronitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oculomotor and pupillomotor quantitative measurements (Experimental): The investigators will assess oculomotor and pupillomotor function at the bedside and quantitatively both in the acute stage (i.e., within the first 5 days after symptom onset on the ward) and again after 3 months at follow-up (in the outpatient center). They will measure visually-triggered saccadic eye movements and pursuit eye movements in the horizontal and vertical plane and assess pupillary responses to light. For comparison with established paradigms, they will also assess spontaneous nystagmus at primary gaze (with/without fixation), vertical ocular alignment on alternating cover test (looking for vertical deviations, termed skew deviation), gaze-evoked nystagmus on lateral gaze (GEN), and the horizontal head-impulse test (hHIT). The investigators will also test hearing. Bedside and quantitative testing will be performed at the same time.
  Interventions: Diagnostic Test: video-oculography

INTERVENTIONS:
Diagnostic Test: video-oculography — All participants will receive quantitative oculomotor and pupillomotor measurements using two different video-oculography devices. Thereby both pursuit eye movements, saccades and pupillary responses to light will be assessed. In addition, there will be a quantitative assessment of the angular vestibulo-ocular reflex (aVOR) by use of video-head-impulse testing and a hearing test.

SUMMARY:
BACKGROUND: A chief complaint of acute vertigo/dizziness is related to about 2.1-7.1% of all emergency department (ED) visits. About 25% of all patients with acute prolonged vertigo meeting diagnostic criteria of AVS (acute vestibular syndrome) suffer from a vertebrobasilar stroke and about 35% of these patients are initially missed. Differentiating dangerous central from more benign peripheral causes of AVS is essential. Subtle oculomotor paradigms such as HINTS (Head-Impulse, Nystagmus, Test-of-Skew) have been shown to detect central causes with high diagnostic accuracy, however, require sufficient training. Thus, identifying other bedside tests that can be reliably performed by frontline providers is essential to reduce misdiagnosis.

WORKING HYPOTHESIS: By using additional oculomotor (saccades, pursuit) and pupillomotor parameters at the bedside or quantitatively, the diagnostic accuracy for distinguishing peripheral from central AVS causes can be further improved, especially in the setting when expertise for applying more sophisticated algorithms (HINTS(+), STANDING) is lacking.

AIM 1: Detecting changes in oculomotor and pupillomotor responses in acutely dizzy patients and characterizing the spectrum of abnormalities in peripheral and central AVS.

AIM 2: Comparing different composite oculomotor-/pupillomotor scores to identify those scores with the highest diagnostic accuracy at the bedside and quantitatively.

AIM 3: Comparing the diagnostic accuracy of bedside and quantitative oculomotor and pupillomotor testing in AVS- identifying potential limitations of bedside testing.

METHODS: To assess oculomotor and pupillomotor responses in patients with peripheral or central AVS and healthy controls (25 participants each) at the bedside and quantitatively by use of a Pioneer research eye tracker (PRET) system and to compare the diagnostic accuracy of individual and composite responses.

EXPECTED VALUE OF THE PROJECT: The proposed project will shed more light on the value of different examination techniques in AVS for distinguishing peripheral from central causes. This is achieved by investigating oculomotor and pupillomotor parameters obtained at the bedside and quantitatively in the acute stage and at follow-up. The insights gained will likely have a direct impact on diagnostic accuracy and thus on future strategies how to evaluate acutely dizzy patients in the ED. Eventually, this may reduce the rate of misdiagnosis and may improve patients' outcome.

DETAILED DESCRIPTION:
A chief complaint of acute vertigo or dizziness is related to about 2.1 to 7.1% of all emergency department (ED) visits, translating to about 4.3 million ED visits in the USA per year. With the differential diagnosis of patients presenting with acute or episodic vertigo / dizziness being very broad and cutting across all specialties, frontline providers and specialists may be overwhelmed by the approach to this symptom. In patients presenting to the ED with vestibular symptoms, life-threatening conditions have been identified in a single study in 23.8% of visits, with 12.5% of all visits related to cerebrovascular events. This emphasizes the need to distinguish between dangerous central and benign, self-limited peripheral vestibular disorders to avoid misdiagnosis. Patients with an acute vestibular syndrome (AVS) have acute-onset, continuous vertigo, dizziness, or unsteadiness lasting days to weeks, usually associated with vomiting, nystagmus, severe postural instability and head movement intolerance . Both patients with stroke and vestibular neuritis can present with an AVS. Approximately 25%±15% of AVS patients will be diagnosed with a stroke, usually in the posterior circulation. Established diagnostic workup in the ED include neurologic assessment, followed usually by CT-based imaging of the brain. Often neurology consultations will be ordered.

For posterior circulation strokes presenting with dizziness frontline misdiagnosis appears common, occurring in roughly 35% of cases. The desire to avoid missing a stroke often triggers brain imaging (computed tomography [CT] and magnetic resonance imaging including diffusion-weighted imaging [MRI-DWI]), laboratory workup and/or electrocardiography. Unfortunately, a recent meta-analysis found that the sensitivity of CT for central causes of dizziness was only 28.5%. Even MRI-DWI in AVS has limited sensitivity, missing about 1 out of 5 vertebrobasilar strokes presenting as an AVS when obtained within the first 24-48 hours after symptom onset. If stroke, the most common central cause of the AVS is missed or delayed, the underlying stroke mechanism goes untreated sometimes resulting in extension of the original infarct or development of a new, larger one.

The evidence base for effective bedside differentiation of inner ear diseases from stroke in patients with acute dizziness and vertigo has grown substantially over time, as emphasized recently. Although useful if present, obvious focal neurologic signs only have a sensitivity of 44% for detecting a central cause of AVS, i.e., more than 50% of strokes will be missed if one were to rely on these findings. Thus, different clinical strategies that emphasize the combined use of targeted neuro-otologic bedside examination techniques, such as the HINTS (Head Impulse, Nystagmus, Test of Skew), HINTS+ (which adds a bedside test of hearing), STANDING or gait/truncal instability (GTI) assessment have been proposed.

Both the HINTS(+) exam and the STANDING algorithm are very good exclusion tests in the hands of trained emergency physicians, non-sub-specialists and neuro-otology / neuro-ophthalmology subspecialists. Ideally, HINTS+ are combined with a graded GTI rating or the STANDING algorithm is used instead. However, absent or inadequate training in performing and interpreting subtle oculomotor findings constitute important limitations, especially in frontline providers. Most ED physicians are not yet familiar with a structured approach to the dizzy patient as e.g. outlined in the TiTrATE approach and HINTS(+) or similar bedside algorithms. While the introduction of quantitative (video oculography - VOG) HINTS to the ED seems promising, increasing the diagnostic accuracy beyond that of neuro-otology experts, this concept is far from being implemented broadly in routine emergency medicine practice.

This emphasizes the need to further improve the approach to the acutely dizzy patient now, focusing on bedside testing that can be reliably applied by untrained frontline providers including emergency physicians or neurology residents also. Brainstem and cerebellar loss of function have been demonstrated to result in dysmetric saccades and saccadic pursuit eye movements. In a previous study, vertical pursuit was saccadic significantly more often in central AVS patients than in peripheral AVS patients (88% vs. 20%, p<0.01). In patients with (dorso)lateral medullary lesions or carotid artery dissection, pupillary abnormalities (Horner syndrome) may be noticed and in midbrain lesions an unilaterally dilated pupil (as part of a third nerve palsy) may be observed, whereas for other acute brainstem or for cerebellar lesions little is known about pupillomotor changes. Testing for both saccadic eye movements (SEM), pursuit eye movements (PEM) and pupillary responses is straight-forward and readily applicable by frontline providers.

In this proposal the investigators will address the question whether by using additional oculomotor (SEM, PEM) and pupillomotor (pupillary constriction to light) parameters at the bedside or quantitatively, the diagnostic accuracy for distinguishing peripheral from central causes in AVS can be further improved or not. This will be especially important in any setting where expertise for applying more sophisticated algorithms such as HINTS(+) or STANDING is lacking.

The risk for this study protocol is minimal (Risk Category A) due to the non-invasive nature of the measurements obtained (video-oculography, audiometry), side-effects anticipated are expected to be mild and transient only (discomfort by wearing the video-oculography device, vertigo or dizziness being more intense during the measurements, mild nausea).

The investigators do not anticipate an impact of "sex and gender" on the parameters measured, but they will assess the presence/absence of gender impact by statistical analysis.

The overriding hypothesis of this proposal is, that by using additional oculomotor (SEM, PEM) and pupillomotor (pupillary constriction to light) parameters at the bedside or quantitatively, the diagnostic accuracy for distinguishing peripheral from central causes in AVS can be further improved, especially in the setting when expertise for applying more sophisticated algorithms such as HINTS(+) or STANDING is lacking. To address this, the investigators will first collect oculomotor, pupillomotor and vestibular responses in AVS patients within the first 5 days after symptom onset, characterizing the spectrum of changes in peripheral and central causes of AVS (Aim 1). The gold standard will be brain MRI including diffusion-weighted imaging (DWI), obtained between 48 hours and 14 days after symptom onset. The investigators will compare different composite oculomotor-/pupillomotor scores to identify those scores with the highest diagnostic accuracy (Aim 2). Furthermore, comparing results retrieved when testing clinically at the bedside and quantitatively will allow the investigators to better understand if changes in SEM, PEM and pupillary responses as measured quantitatively will also be perceived by the examiner at the bedside (Aim 3). This will be critical to judge the value and thus the priority for testing these parameters at the bedside.

ELIGIBILITY:
Inclusion Criteria:

* Patient groups

  * patients presenting with an AVS (peripheral or central), with symptom duration of 5 days or less
  * being able to receive brain MRI
* All groups:

  * Being able to give informed consent as documented by signature
  * Age 18 years or above

Exclusion Criteria:

* Aged less than 18 years.
* Pregnant or lactating women
* Inability or contraindications to undergo the investigated intervention (including brain MRI in the patient groups),
* Clinically significant concomitant diseases such neurodegenerative disorders (e.g. Alzheimer's disease, Parkinson's disease)
* Pre-existing peripheral-vestibular / central-vestibular deficits
* History of brainstem / cerebellar stroke
* Pre-existing or acute severe visual loss
* Pre-existing severe hearing loss.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, aphasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy in visually-guided saccades in patients with AVS | Two sessions will be recorded 3 months apart. For patients, session 1 will be obtained within 5 days after symptom onset
  As the primary end point of our interventional study, the investigators selected the diagnostic accuracy of horizontal and vertical visually-guided saccades (calculated gain, looking for hypermetria and hypometria) in patients with either central or peripheral AVS (time points: acutely, at 3-month follow-up) and in comparison to healthy controls. Differences in quantitative saccade responses in the distinct study groups will support their future use in the acute evaluation of such patients in the ED and will help guide the ED physician in the selection of tests and their interpretation. In the secondary end points (see below), the investigators will also address to which extent the combination of quantitative oculomotor parameters may improve diagnostic accuracy.

SECONDARY OUTCOMES:
Diagnostic accuracy for HINTS+ vs. brain MRI-DWI for detecting central AVS cases | One measurement in all AVS patients within 5 days of symptom-onset
  Here the investigators will compare the diagnostic accuracy (sensitivity, specificity, NLR, PLR) of the HINTS+ score vs. brain MRI-DWI for detecting central (mostly ischemic) AVS causes. This comparison is thus between a bedside clinical score and imaging.
Diagnostic accuracy in pursuit eye movements in AVS patients for predicting a central origin | Two sessions will be recorded 3 months apart. For patients, session 1 will be obtained within 5 days after symptom onset
  For this secondary aim, quantitative pursuit eye movement measurements (both in the horizontal and vertical) plane obtained within 5 days after symptom onset in the AVS patients are obtained and their diagnostic value for distinguishing between peripheral and central AVS cases is evaluated. For comparison, the same measurements will also be obtained in healthy controls.
Pupillary constriction to light (gain) | Two sessions will be recorded 3 months apart. For patients, session 1 will be obtained within 5 days after symptom onset
  Pupillary constriction to bright light is assessed by use of the PRET video-oculography device, comparing findings in AVS patients and healthy controls. Diagnostic accuracy for detecting central AVS cases will be determined based on the pupillary response.
Diagnostic accuracy of a combined oculomotor-pupillomotor score vs. HINTS+ | Two sessions will be recorded 3 months apart. For patients, session 1 will be obtained within 5 days after symptom onset
  Here a combined oculomotor-pupillomotor score (gain of saccades, gain of pursuit and pupillary gain) is compared agains an established bedside evaluation (HINTS+). Specifically, the diagnostic accuracy of both scores for detecting an underlying central cause of the patient's AVS is calculated.
aVOR gain of both horizontal and vertical semicircular canals | Two sessions will be recorded 3 months apart. For patients, session 1 will be obtained within 5 days after symptom onset
  Here the gain of the angular vestibulo-ocular reflex (aVOR) responses for all six semicircular canals (as assessed by use of video-head-impulse testing) are compared for both peripheral and central AVS patients and healthy controls. Reduced aVOR gains are anticipated for all patients with peripheral AVS and in about 20% of patients with central AVS.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander A Tarnutzer, MD, Principal Investigator — Neurology, Cantonal Hospital of Baden, Baden, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication

REFERENCES:
- [Background] Cnyrim CD, Newman-Toker D, Karch C, Brandt T, Strupp M. Bedside differentiation of vestibular neuritis from central "vestibular pseudoneuritis". J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):458-60. doi: 10.1136/jnnp.2007.123596. PMID 18344397
- [Background] Carmona S, Martinez C, Zalazar G, Moro M, Batuecas-Caletrio A, Luis L, Gordon C. The Diagnostic Accuracy of Truncal Ataxia and HINTS as Cardinal Signs for Acute Vestibular Syndrome. Front Neurol. 2016 Aug 8;7:125. doi: 10.3389/fneur.2016.00125. eCollection 2016. PMID 27551274
- [Background] Bogousslavsky J, Meienberg O. Eye-movement disorders in brain-stem and cerebellar stroke. Arch Neurol. 1987 Feb;44(2):141-8. doi: 10.1001/archneur.1987.00520140013011. PMID 3545158
- [Background] Vanni S, Nazerian P, Casati C, Moroni F, Risso M, Ottaviani M, Pecci R, Pepe G, Vannucchi P, Grifoni S. Can emergency physicians accurately and reliably assess acute vertigo in the emergency department? Emerg Med Australas. 2015 Apr;27(2):126-31. doi: 10.1111/1742-6723.12372. Epub 2015 Mar 10. PMID 25756710
- [Background] Tarnutzer AA, Gold D, Wang Z, Robinson KA, Kattah JC, Mantokoudis G, Saber Tehrani AS, Zee DS, Edlow JA, Newman-Toker DE. Impact of Clinician Training Background and Stroke Location on Bedside Diagnostic Test Accuracy in the Acute Vestibular Syndrome - A Meta-Analysis. Ann Neurol. 2023 Aug;94(2):295-308. doi: 10.1002/ana.26661. Epub 2023 Apr 27. PMID 37038843
- [Background] Tarnutzer AA, Berkowitz AL, Robinson KA, Hsieh YH, Newman-Toker DE. Does my dizzy patient have a stroke? A systematic review of bedside diagnosis in acute vestibular syndrome. CMAJ. 2011 Jun 14;183(9):E571-92. doi: 10.1503/cmaj.100174. Epub 2011 May 16. No abstract available. PMID 21576300
- [Background] Shah VP, Oliveira J E Silva L, Farah W, Seisa M, Kara Balla A, Christensen A, Farah M, Hasan B, Bellolio F, Murad MH. Diagnostic accuracy of neuroimaging in emergency department patients with acute vertigo or dizziness: A systematic review and meta-analysis for the guidelines for reasonable and appropriate care in the emergency department. Acad Emerg Med. 2023 May;30(5):517-530. doi: 10.1111/acem.14561. Epub 2022 Aug 17. PMID 35876220
- [Background] Newman-Toker DE, Kerber KA, Hsieh YH, Pula JH, Omron R, Saber Tehrani AS, Mantokoudis G, Hanley DF, Zee DS, Kattah JC. HINTS outperforms ABCD2 to screen for stroke in acute continuous vertigo and dizziness. Acad Emerg Med. 2013 Oct;20(10):986-96. doi: 10.1111/acem.12223. PMID 24127701
- [Background] Newman-Toker DE, Edlow JA. TiTrATE: A Novel, Evidence-Based Approach to Diagnosing Acute Dizziness and Vertigo. Neurol Clin. 2015 Aug;33(3):577-99, viii. doi: 10.1016/j.ncl.2015.04.011. PMID 26231273
- [Background] Kattah JC, Talkad AV, Wang DZ, Hsieh YH, Newman-Toker DE. HINTS to diagnose stroke in the acute vestibular syndrome: three-step bedside oculomotor examination more sensitive than early MRI diffusion-weighted imaging. Stroke. 2009 Nov;40(11):3504-10. doi: 10.1161/STROKEAHA.109.551234. Epub 2009 Sep 17. PMID 19762709
- [Background] Saber Tehrani AS, Coughlan D, Hsieh YH, Mantokoudis G, Korley FK, Kerber KA, Frick KD, Newman-Toker DE. Rising annual costs of dizziness presentations to U.S. emergency departments. Acad Emerg Med. 2013 Jul;20(7):689-96. doi: 10.1111/acem.12168. PMID 23859582
- [Background] Newman-Toker DE, McDonald KM, Meltzer DO. How much diagnostic safety can we afford, and how should we decide? A health economics perspective. BMJ Qual Saf. 2013 Oct;22 Suppl 2(Suppl 2):ii11-ii20. doi: 10.1136/bmjqs-2012-001616. No abstract available. PMID 24048914
- [Background] Newman-Toker DE, Hsieh YH, Camargo CA Jr, Pelletier AJ, Butchy GT, Edlow JA. Spectrum of dizziness visits to US emergency departments: cross-sectional analysis from a nationally representative sample. Mayo Clin Proc. 2008 Jul;83(7):765-75. doi: 10.4065/83.7.765. PMID 18613993
- [Background] Goeldlin M, Gaschen J, Kammer C, Comolli L, Bernasconi CA, Spiegel R, Bassetti CL, Exadaktylos AK, Lehmann B, Mantokoudis G, Kalla R, Fischer U. Frequency, aetiology, and impact of vestibular symptoms in the emergency department: a neglected red flag. J Neurol. 2019 Dec;266(12):3076-3086. doi: 10.1007/s00415-019-09525-4. Epub 2019 Sep 17. PMID 31531764
- [Background] Ljunggren M, Persson J, Salzer J. Dizziness and the Acute Vestibular Syndrome at the Emergency Department: A Population-Based Descriptive Study. Eur Neurol. 2018;79(1-2):5-12. doi: 10.1159/000481982. Epub 2017 Nov 13. PMID 29131011
- [Background] Kerber KA, Meurer WJ, West BT, Fendrick AM. Dizziness presentations in U.S. emergency departments, 1995-2004. Acad Emerg Med. 2008 Aug;15(8):744-50. doi: 10.1111/j.1553-2712.2008.00189.x. Epub 2008 Jul 14. PMID 18638027
- [Background] Kerber KA, Brown DL, Lisabeth LD, Smith MA, Morgenstern LB. Stroke among patients with dizziness, vertigo, and imbalance in the emergency department: a population-based study. Stroke. 2006 Oct;37(10):2484-7. doi: 10.1161/01.STR.0000240329.48263.0d. Epub 2006 Aug 31. PMID 16946161